CLINICAL TRIAL: NCT03340779
Title: Norepinephrine vs Norepinephrine and Dobutamine in Cardiogenic Shock : a Randomised, Opened, Cross-over Study. Heart SHOCK-NORDOB Study
Brief Title: Norepinephrine vs Norepinephrine and Dobutamine in Cardiogenic Shock
Acronym: SHOCK-NORDOB
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2017-001270-41
Record Dates: First submitted 2017-09-20; First posted 2017-11-14 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-09

CONDITIONS: Cardiogenic Shock
Keywords: Norepinephrine; Dobutamine; Shock
MeSH Terms: conditions — Shock, Cardiogenic; Shock | interventions — Norepinephrine; Dobutamine

STUDY DESIGN:
Intervention Model Description: 3 first hours : strategy 1, norepinephrine alone with increased dose or norepinephrine + dobutamine 0.5 hour : wash-out (decrease of norepinephrine dose or weaning of dobutamine) 3 last hours : strategy 2, crossover, norepinephrine alone with increased dose or norepinephrine + dobutamine
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Norepinephrine alone (Experimental): Administration of norepinephrine with increasing dose
  Interventions: Drug: Norepinephrine
- Norepinephrine plus Dobutamine (Active Comparator): Administration of norepinephrine and dobutamine
  Interventions: Drug: Norepinephrine

INTERVENTIONS:
Drug: Norepinephrine — After obtention of a mean arterial pressure (MAP) of 65 mmHg with infusion of norepinephrine, patients with cardiogenic shock receive for 3 hours either increasing doses of norepinephrine (with a maximal MAP of 85 mmHg) or dobutamine. There is a wash-out phase of 30 minutes (decrease of norepinephrine dose or weaning of dobutamine). The third phase of the study is the administration of the comparator treatment during 3 hours. After the 6.5 hours of the study, the hemodynamic management is up to the physician.
  Other Names: Dobutamine

SUMMARY:
Cardiogenic shock is a frequent cause of admission and death in the intensive care unit.

Mortality is about 50%. Once the etiologic treatment has been done, for instance coronary revascularization, management of the shock state is the cornerstone of the treatment. Norepinephrine is the first-line vasopressor therapy because of its minor effect on heart rhythm. Morever norepinephrine is a inotrope. In a previous study, we demonstrated that increasing the norepinephrine dose increases cardiac index, cardiac power index, SVO2 and tissue perfusion without acceleration of heart rate. Nevertheless, dobutamine remains the first-line inotropic treatment. Dobutamine has a positive chronotropic effect that might cause higher myocardial oxygen consumption. As a result, combination of vasopressor / inotrope is still controversial.

The aim of this study was to compare hemodynamics and metabolics effects of 2 treatments strategies (norepinephrine dose increasing or addition of dobutamine) in patients with cardiogenic shock and optimised blood pressure level (MAP≥65 mmHg) under norepinephrine treatment.

The secondary objectives were :

* To evaluate the efficacy of the treatments on micro- and macrocirculation parameters
* To evaluate the tolerance of the treatments
* To evaluate the dose and the admistration's kinetics of the treatments

ELIGIBILITY:
Inclusion Criteria:

* Patients with cardiogenic shock (ischemic, rythmic, valvular) defined : by cardiac index (CI) < 2,2 L/min/m² or CI < 2,5 L/min/m² under vasopressor/inotropic treatment and organ hypoperfusion signs : mottles, capillary refill time , urine output < 0,5 mL/kg/hour during at least one hour ou renal replacement therapy, consciouness impairment, pulmonary oedema, hyperlactatemia (> 2 mmoL/L)
* Mean arterial pressure > 65 mmHg under norepinephrine treatment
* Patients with social coverage

Exclusion Criteria:

* < 18 years old
* Pregnancy
* Inclusion in other drug study
* Poisonings with cardiotoxicants
* Patient with intra-aortic ballon pump, extracorporeal life support
* Patient under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-01-15 (Estimated); Primary Completion 2019-11-01 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Obtention of a optimal cardiac output | Hour 0 (H0), Hour 1, Hour 3, Hour 3.5, Hour 4,5, Hour 5.5, Hour 6.5
  Measure of increase of cardiac index > 15% (L/min/m²), increase of organ perfusion assessed by : lactate clearance > 15% (mmoL/L), decrease of mottling (decrease of 2 points of Mottling score), increase of musculaire oxygen saturation measured by NIRS > 15% (rSo2%), increase of urine output > 50% (mL/h), increase of SVcO2 > 15%(%)
  Evaluation of occurence of side effects :
  Increase of heart rate > 15% (bpm) , increase of oxygen consumption evaluated by decrease of ratio mean arterial pressure / heart rate > 15% (Buffington ratio).
  The primary endpoint is defined by the presence of 2 efficacy criterias without any side effects.

SECONDARY OUTCOMES:
Change in hemodynamic parameters | Hour 0, Hour 1, Hour 3, Hour 3.5, Hour 4,5, Hour 5.5, Hour 6.5
  Measure of heart rate (bpm),
Occurence of arrythmia | Hour 0, Hour 1, Hour 3, Hour 3.5, Hour 4,5, Hour 5.5, Hour 6.5
  Notification of atrial arrythmia
Change in hemodynamic parameters | Hour 0, Hour 1, Hour 3, Hour 3.5, Hour 4,5, Hour 5.5, Hour 6.5
  Cumulated dose of catecholamines
All-cause mortality | Day 28
  Mortality
Change in hemodynamic parameters | Hour 0, Hour 1, Hour 3, Hour 3.5, Hour 4,5, Hour 5.5, Hour 6.5
  Arterial blood pressure (mmHg)
Change in metabolic parameters | Hour 0, Hour 1, Hour 3, Hour 3.5, Hour 4,5, Hour 5.5, Hour 6.5
  SVcO2 (%)
Change in metabolic parameters | Hour 0, Hour 1, Hour 3, Hour 3.5, Hour 4,5, Hour 5.5, Hour 6.5
  Lactate clearance (mmol/L)
Change in metabolic parameters | Hour 0, Hour 1, Hour 3, Hour 3.5, Hour 4,5, Hour 5.5, Hour 6.5
  Muscular oxygen saturation (%)
Change in metabolic parameters | Hour 0, Hour 1, Hour 3, Hour 3.5, Hour 4,5, Hour 5.5, Hour 6.5
  Urine output (mL/h)
Change in metabolic parameters | Hour 0, Hour 1, Hour 3, Hour 3.5, Hour 4,5, Hour 5.5, Hour 6.5
  Mottle (mottle score)
Occurence of arrythmia | Hour 0, Hour 1, Hour 3, Hour 3.5, Hour 4,5, Hour 5.5, Hour 6.5
  Notification of ventricular arrythmia

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Nancy-Brabois, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No